CLINICAL TRIAL: NCT01326975
Title: Effects of Continuous Positive Airway Pressure (CPAP) Delivered by High Flow Nasal Cannula Versus Nasal Continuous Positive Airway Pressure on the Diaphragm Electrical Activity in Very Low Birth Weight Preterm Infants
Brief Title: Effect of Continuous Positive Airway Pressure Delivered by Two Different Modalities on Breathing Pattern in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 254-2010
Record Dates: First submitted 2011-03-23; First posted 2011-03-31 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Continuous Positive Airway Pressure
Keywords: infant, premature; infant, very low birth weight; diaphragm; apnea; continuous positive airway pressure
MeSH Terms: conditions — Premature Birth; Apnea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- EAdi 1: babies in this group will first receive CPAP through IF-CPAP for 30 minutes. After another 45 minutes, they will be switched to HFNC for 30 minutes. EAdi will be recorded for the last 15 minutes of each 30 minutes period.
- EAdi 2: babies in this group will first receive CPAP through HFNC for 30 minutes. After another 45 minutes, they will be switched to IF-CPAP for 30 minutes. EAdi will be recorded for the last 15 minutes of each 30 minutes period.

SUMMARY:
In this study, the investigators want to observe how continuous positive airway pressure delivered by two different modalities affects breathing pattern in small preterm infants. Using a specialized feeding tube in the stomach, the investigators can measure and compare how the diaphragm (a large breathing muscle) might be affected by those two modalities.

DETAILED DESCRIPTION:
Many preterm very low birth weight infants require continuous positive airway pressure(CPAP) for breathing support because of lung immaturity. CPAP can be delivered by the infant flow(TM) device which is well studied. Prolonged use of nasal prongs CPAP has been shown to cause discomfort and, rarely, nasal injury leading to long term disfigurement. On the other hand, High flow nasal cannula (HFNC) ,which is another modality of delivering CPAP, creates less pressure on the nose and less disfiguring effect but previous research showed that the use of HFNC may be less effective than IF-CPAP in providing breathing support in these infants.

We plan to study 10 stable preterm infants born less than 32 weeks' gestation and 1.5 kilograms at birth after being stable for at least 48hours on IF-CPAP. babies will be randomized to start on IF-CPAP or HFNC for 30 minutes. After 45 minutes of adaptation, baby will be switched to the other modality for another 30 minutes. By inserting a specialized feeding tube with sensors into the stomach, we can measure the electrical activity of the diaphragm (EAdi). By analysing EAdi with each modality of delivering CPAP, we want to directly assess how HFNC affects breathing compared to IF-CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Birth weights ≤ 1500g
* Gestational age less than 32 week
* Stable on nasal continuous positive airway pressure (CPAP) of 5-6cmH20 support for at least 48 hours
* Treated with methylxanthines for apnea of prematurity
* In less than 35% oxygen

Exclusion Criteria:

* Congenital and acquired problem of the gastrointestinal tract
* Phrenic nerve injury and/or diaphragm paralysis
* Esophageal perforation/tracheoesophageal fistula
* Congenital/acquired neurological deficit and/or seizures
* Hemodynamic instability
* Congenital heart disease (including symptomatic patent ductus arteriosus)
* Undergoing treatment for sepsis or pneumonia
* Use of muscle relaxants, narcotic analgesics, or gastric motility agents
* Congenital anomalies of respiratory tract (e.g. CCAM)
* Infants requiring more than 35% oxygen
* Infants with facial anomalies
* Infants with pneumothorax and/or pneumomediatinum
* Infants in the immediate postoperative period
* Infants with significant gastric residues and vomiting

Ages: 2 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: clinically stable preterm infants with birth weight less than 1.5 kilograms and gestational age less than 32 weeks admitted to the neonatal intensive care unit at Sunnybrook Health Sciences centre on nasal continuos positive airway pressure(CPAP) of 5-6 cmH2O support for at least 48 hours, treated with Methylxanthines for apnea of prematurity and in less than 35% oxygen.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The difference in the tonic EAdi between IF-CPAP and HFNC . | During the 4-hour study period.
  Patients will be randomized in two groups, one group will start on IF-CPAP for 30 minutes. After another 45 minutes, this group will be switched to HFNC for another 30 minutes. The other group will start on HFNC and then switched to IF-CPAP. EAdi will be analyzed in the last 15 minutes of each 30 minutes period.

SECONDARY OUTCOMES:
Difference in the number of apnea episodes (breathing pauses) on EAdi recorded with each modality. | During the 4-hour study period.
Difference in episodes of clinically significant apnea with HFNC and IF-CPAP. | During the 4-hour study period.
Indices of respiratory muscle effort (inspiratory and expiratory) will be calculated from Edi waveform. | During the 4-hour study period.
  These indices include the phasic Edi to the peak, mean inspiratory Edi, Edi-time product, post inspiratory activity and all neural timings.

CONTACTS AND LOCATIONS:
Overall Officials: Nehad Nasef, M.B.B.Ch, Principal Investigator — Sunnybrook Health Sciences Centre; Maureen Reilly, RRT, Principal Investigator — Sunnybrook Health Sciences Centre; Patti Schurr, RN(EC), Principal Investigator — Sunnybrook Health Sciences Centre; Michael Dunn, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Jennifer Beck, Ph.D., Principal Investigator — Unity Health Toronto; Eugene Ng, MD, Study Director — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada